CLINICAL TRIAL: NCT02945488
Title: Exercise and Nutrition as Treatment Alternatives in Women With Inflammatory Bowel Disease During Preconception: Saskatchewan Multidisciplinary Inflammatory Bowel Diseases Clinic (MDIBDC)
Brief Title: Exercise and Nutrition in IBD & Preconception
Acronym: IBDPreconcep
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Saskatchewan Health Research Foundation (Other); Crohn's and Colitis Canada (Other)
Responsible Party: Principal Investigator, Sharyle Fowler, M.D., University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-132
Record Dates: First submitted 2016-09-27; First posted 2016-10-26 (Estimated); Last update posted 2018-06-13 (Actual); Status verified 2018-06

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Exercise and dietary plan (Experimental): Combination cardiovascular and resistance training and Mediterranean dietary plan
  Interventions: Other: Exercise; Other: Dietary plan
- Exercise and no dietary plan (Experimental): Combination cardiovascular and resistance training and participants regular diet (control diet)
  Interventions: Other: Exercise
- Stretching and dietary plan (Experimental): Flexibility training (control exercise) and Mediterranean dietary plan
  Interventions: Other: Dietary plan; Other: Stretching
- Stretching and no dietary plan (Active Comparator): Flexibility training (control exercise) and participants regular diet (control diet)
  Interventions: Other: Stretching

INTERVENTIONS:
Other: Exercise — Exercise intervention will entail 30 minutes of moderate intensity cardiovascular training 3 days/week and full body resistance training 2 days/week (supervised). Cardiovascular training will entail any weight-bearing activity that would achieve target heart rate, such as walking, jogging, stair climbing, dancing, etc. Resistance training will entail 2-3 sets of 8-12 repetitions of exercises targeting all major muscle groups with an external load applied, such as a dumbbell, barbell, medicine ball, etc.
  Arms: Exercise and dietary plan; Exercise and no dietary plan
Other: Dietary plan — Mediterranean dietary plan, which contains foods, such as fish, vegetables, nuts, and oils, which are anti-inflammatory in nature.
  Arms: Exercise and dietary plan; Stretching and dietary plan
Other: Stretching — Stretching intervention will entail 30 minutes of flexibility training 3 days/week of stretches targeting all major muscle groups held for 20-30 seconds.
  Arms: Stretching and dietary plan; Stretching and no dietary plan

SUMMARY:
The objectives are to: 1) Assess the independent and synergistic efficacy of exercise and nutrition interventions to manage major symptomatic concerns of inflammatory bowel diseases (IBD), 2) Assess the independent and synergistic efficacy of exercise and nutrition to mitigate inflammation in IBD, and 3) Assess the feasibility of such an intervention in preconception women with IBD. The investigators hypothesize that the combination of anti-inflammatory exercise and nutritional interventions will have a synergistic effect on managing major symptomatic concerns associated with IBD, reducing inflammation, and improving fertility status in preconception women with IBD, as compared to either intervention independently.

DETAILED DESCRIPTION:
Potential participants will be recruited from the Preconception and Pregnancy Clinic recently established within the Saskatchewan Multidisciplinary Inflammatory Bowel Disease Clinic [MDIBDC]. Eligible participants will be randomized [stratified] to one of four groups: 1) Exercise and dietary plan, 2) Exercise and no dietary plan, 3) Stretching [placebo exercise] and dietary plan, 4) Stretching and no dietary plan. Participants will be assessed at baseline, midway [3 months], and post-intervention [6 months] for indications of disease activity, quality of life, fertility status, and bone health.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Confirmed diagnosis of Inflammatory Bowel Disease
* Child-bearing age

Exclusion Criteria:

* Currently following a Mediterranean diet
* Currently performing resistance training on a regular basis (within the past 6 months)
* Failed Physical Activity Readiness Questionnaire-Plus (PAR-Q+).
* Past ileal pouch anal anastomosis
* Unstable or uncontrolled cardiovascular, pulmonary, hepatic, renal, gastrointestinal, or other medical disorder that, in the opinion of the investigator, would confound the study results or compromise subject safety

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Inflammatory Bowel Disease Questionnaire score | Baseline, 3 months, and 6 months
  Inflammatory Bowel Disease Questionnaire (score on a scale); measures quality of life

SECONDARY OUTCOMES:
Change from Baseline Interleukin-6 | Baseline, 3 months, and 6 months
  Serum Interleukin-6 (pg/mL); measures inflammation
Change from Baseline in Follicle Stimulating Hormone | Baseline, 3 months, and 6 months
  Serum Follicle Stimulating Hormone (mIU/ml); measures fertility status
Change from Baseline in Leisure Time Physical Activity Questionnaire score | Baseline, 3 months, and 6 months
  Leisure Time Physical Activity Questionnaire (arbitrary score); measures physical activity levels outside intervention
Change from Baseline in Estradiol | Baseline, 3 months, and 6 months
  Serum estradiol (pg/mL); measures fertility status
Change from Baseline in Total Body Lean Mass | Baseline, 3 months, and 6 months
  Total body lean mass (grams) via dual energy x-ray absorptiometry scan; measures body composition
Change from Baseline in Total Body Fat Mass | Baseline, 3 months, and 6 months
  Total body fat mass (grams) via dual energy x-ray absorptiometry scan; measures body composition
Change from Baseline in Body Composition | Baseline, 3 months, and 6 months
  Body fat percentage (%) via dual energy x-ray absorptiometry scan; measures body composition
Change from Baseline in Femoral Neck Bone Mineral Density | Baseline, 3 months, and 6 months
  Femoral neck bone mineral density (g/cm^2) via dual energy x-ray absorptiometry scan; measures bone health
Change from Baseline in Total Body Bone Mineral Density | Baseline, 3 months, and 6 months
  Total body bone mineral density (g/cm^2) via dual energy x-ray absorptiometry scan; measure bone health
Change from Baseline in Harvey Bradshaw Index | Baseline, 3 months, and 6 months
  Harvey Bradshaw Index for Crohn's disease (score on a scale); measures clinical disease activity
Change from Baseline in partial Mayo Score | Baseline, 3 months, and 6 months
  Partial Mayo Score for ulcerative colitis (score on a scale); measures clinical disease activity
Change from Baseline Fecal Calprotectin | Baseline, 3 months, and 6 months
  Fecal calprotectin (mg/kg); measures clinical disease activity
Change from Baseline Protein Consumption | Baseline, 3 months, and 6 months
  Food Frequency Questionnaire average protein consumption per day (grams); measures nutritional status
Change from Baseline Carbohydrate Consumption | Baseline, 3 months, and 6 months
  Food Frequency Questionnaire average carbohydrate consumption per day (grams); measures nutritional status
Change from Baseline Fat Consumption | Baseline, 3 months, and 6 months
  Food Frequency Questionnaire average fat consumption per day (grams); measures nutritional status
Change from Baseline EuroQol Five Dimensions Questionnaire (EQ-5D) score | Baseline, 3 months, and 6 months
  The EQ-5D (score on a scale); measures quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Sharyle Fowler, MD, Principal Investigator — University of Saskatchewan
Locations (1):
- Royal University Hospital, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No